CLINICAL TRIAL: NCT01495975
Title: Impact of a Web-based Diabetes Transitions Tool Kit on Post-Hospitalization Glycemic Control
Brief Title: Impact of a Diabetes Transitions Tool Kit on Post-Hospitalization Glycemic Control
Acronym: DTTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Wexler, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Deborah Wexler, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011p-001573; 5K23DK080228-05 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2011-12-20 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Hospitalization; Patient Discharge
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual care for diabetes in the 1 month after discharge.
- Diabetes Transitions Tool Kit (Experimental): Remote glucose monitoring and a web-based patient-provider communication portal, the Diabetes Transitions Toolkit (DTTK), in the 1 month after discharge.
  Interventions: Other: Diabetes Transitions Tool Kit

INTERVENTIONS:
Other: Diabetes Transitions Tool Kit — Access to a remote glucose monitoring and a web-based patient-provider communication portal, the Diabetes Transitions Toolkit (DTTK), for the month after discharge.
  Arms: Diabetes Transitions Tool Kit

SUMMARY:
The goal of this research is to evaluate the impact and feasibility of using web-based patient-provider communication and a remote glucose monitoring tool to improve post-hospitalization glycemic control and patient self-care. The investigators hypothesize that providing patients this web-based tool over a 4-week period after discharge to home will result in more effective glycemic control compared to usual care, and that patients with access to the "tool kit" will have a trend towards improved diabetes self-management and less diabetes-related distress.

DETAILED DESCRIPTION:
Diabetes affects 12-25% of all hospitalized adult patients, and 30% of hospitalized diabetes patients have one or more readmissions within one year. While glycemic control is rarely the primary reason for admission, poor glycemic control has been associated with increased rates of hospitalization and worse clinical outcomes, including infections, poor wound healing, and death. Hospitalization has been proposed as a "teachable moment" for patients with diabetes, as they have intensive contact with a full range of expert clinicians, but the effects of changes implemented during hospitalization after discharge are poorly studied.

The objective of this study is to conduct a randomized controlled trial to test a novel approach to diabetes management in the transition from inpatient to outpatient care. We will assign 40 hospitalized adult patients with type 2 diabetes to usual care or access to a web-based patient-provider communication and remote glucose monitoring tool ("Diabetes Transitions Tool Kit"). Our aims are to evaluate feasibility of implementation of the tool as well as impact on post-discharge glycemic control, diabetes-related self-care and distress. We hypothesize that providing patients this web-based tool over a 4-week period after discharge to home will result in more effective glycemic control compared to usual care, and that patients with access to the "tool kit" will have a trend towards improved diabetes self-management and less diabetes-related distress. Feasibility and preliminary data from this pilot study will be the foundation for larger-scale interventions that may ultimately improve the delivery of diabetes care in the transition from hospital to home.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* English speaking and able to read English
* Diagnosis of type 2 diabetes (new and pre-existing)
* Hospital admission with endocrinology or inpatient diabetes management consult
* On insulin during hospitalization with plan for continuation upon discharge.
* Discharge planned for home.
* Access to the internet and an active email account throughout the 6-week study period.

Exclusion Criteria:

* Inability to connect to, navigate, and utilize the web-based system, or designate someone who is capable of using the system.
* No identifiable outpatient healthcare provider.
* Pregnancy, ruled out by urine hCG test after consent is obtained in all women who continue to have menstrual cycles.
* End-stage liver disease with prothrombin time >15 seconds and albumin <3 mg/dL.
* Hypoglycemia unawareness: patient lacks sensation of common signs of blood glucose <60 mg/dL (tachycardia, diaphoresis, hunger, confusion, fatigue).
* Projected survival <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Wei, MD, Principal Investigator — Massachusetts General Hospital; Deborah J Wexler, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Diabetes Transitions Tool Kit
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Diabetes Transitions Tool Kit | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 52 (14) | 54 (16) | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 11 | 9 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 8 | 16
  Hispanic | 1 | 3 | 4
  Other | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Average HbA1c [Mean (Standard Deviation); unit: %] | 10.2 (2.4) | 10.5 (1.9) | 10.3 (2.2)
Average glycated albumin [Mean (Standard Deviation); unit: %] | 30 (10) | 26 (7) | 28 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Mean patient-day weighted glucose (from glucometer downloads) over the 30 days after discharge
Time Frame: 1 month from discharge
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Diabetes Transitions Tool Kit
Number analyzed (Participants) | 14 | 14
mg/dL | 144 (34) | 172 (41)

2. Secondary Outcome: Diabetes Distress
Description: Measured by the Problem Areas in Diabetes (PAID) Questionnaire
Time Frame: 1 month from discharge
Reporting Status: Not Posted

3. Secondary Outcome: Diabetes Self-Management
Time Frame: 1 month from discharge
Reporting Status: Not Posted

4. Secondary Outcome: Unplanned Readmission or ED Visit
Description: Unplanned readmission to any hospital within 30 days of discharge. Emergency department admission to any hospital within 30 days of discharge.
Time Frame: 1 month after discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Monthly
Arm/Group | Usual Care | Diabetes Transitions Tool Kit
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No